CLINICAL TRIAL: NCT02882386
Title: Does Native Whey Induce Greater Blood Leucine Concentrations Than Other Whey Protein Supplements and Milk: A Randomized Controlled Trial?
Brief Title: Amino Acid Kinetics in Blood After Consuming Different Milk Protein Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Arkansas Children's Hospital Research Institute (Other); Tine (Industry)
Responsible Party: Principal Investigator, Havard Hamarsland, PhD student, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NorwegianSSS
Record Dates: First submitted 2016-08-16; First posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Milk 1% (Placebo Comparator): Participants performed a bout of strength training and consumed 636 ml of a protein supplement
  Interventions: Other: Strength Training; Dietary Supplement: Milk 1%
- Whey protein concentrate 80 (WPC-80) (Experimental): Participants performed a bout of strength training and consumed 636 ml of a protein supplement
  Interventions: Other: Strength Training; Dietary Supplement: Whey protein concentrate 80 (WPC-80)
- Microparticulated whey (Experimental): Participants performed a bout of strength training and consumed 636 ml of a protein supplement
  Interventions: Other: Strength Training; Dietary Supplement: Microparticulated whey
- Hydrolyzed whey (Experimental): Participants performed a bout of strength training and consumed 636 ml of a protein supplement
  Interventions: Other: Strength Training; Dietary Supplement: Hydrolyzed whey
- Native whey (Experimental): Participants performed a bout of strength training and consumed 636 ml of a protein supplement
  Interventions: Other: Strength Training; Dietary Supplement: Native whey

INTERVENTIONS:
Other: Strength Training
Dietary Supplement: Milk 1%
  Other Names: Protein supplementation
  Arms: Milk 1%
Dietary Supplement: Whey protein concentrate 80 (WPC-80)
  Other Names: Protein supplementation
  Arms: Whey protein concentrate 80 (WPC-80)
Dietary Supplement: Microparticulated whey
  Other Names: Protein supplementation
  Arms: Microparticulated whey
Dietary Supplement: Hydrolyzed whey
  Other Names: Protein supplementation
  Arms: Hydrolyzed whey
Dietary Supplement: Native whey
  Other Names: Protein supplementation
  Arms: Native whey

SUMMARY:
The aim of this study is to investigate the amino acid kinetics in blood after a bout of strength training and ingestion of different milk protein supplements (native whey, whey protein concentrate 80, hydrolysed whey, microparticulated whey and milk) The investigators hypothesize that native whey will give a faster and higher rise in blood concentrations of leucine compared to the other milk protein supplements.

DETAILED DESCRIPTION:
Increasing or maintaining muscle mass is of great importance for populations ranging from athletes to patients and elderly. Resistance exercise and protein ingestion are two of the most potent stimulators of muscle protein synthesis. Both the physical characteristic of proteins (e.g. different digestion rates of whey and casein) and the amino acid composition, affects the potential of a certain protein to stimulate muscle protein synthesis. Given its superior ability to rapidly increase blood leucine concentrations to high levels, whey is often considered the most potent protein source to stimulate muscle protein synthesis. Native whey protein is produced by filtration of unprocessed milk. Consequently, native whey has different characteristics than WPC-80, which is exposed to heating and acidification. Because of the direct filtration of unprocessed milk, native whey is a more intact protein compared with WPC-80. Of special interest is the higher amounts of leucine in native whey.

The aim of this double-blinded randomized 5-arm cross-over study is to compare amino acid kinetics in blood after a bout of strength training and ingestion of 20 grams of high quality, but distinct, dairy protein supplements (native whey, whey protein concentrate 80, hydrolysed whey, microparticulated whey and milk). Furthermore, the investigators investigate whether differences in amino acid kinetics affect acute blood glucose and urea response, as well as recovery of muscle function after a bout of strength training.

The investigators hypothesize that native whey will give a faster and higher rise in blood concentrations of leucine compared to the other protein supplements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy in the sense that they can conduct training and testing
* Able to understand Norwegian language written and oral

Exclusion Criteria:

* Diseases or injuries contraindicating participation
* Use of dietary supplements (e.g. proteins, vitamins and creatine)
* Lactose intolerance
* Allergy to milk
* Allergy towards local anesthetics (xylocain)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Plasma amino acid concentration change from baseline | Blood collected at 0, 30, 45, 60, 90 and 120 min after consumption of protein supplements

SECONDARY OUTCOMES:
Serum glucose change from baseline | Blood collected at 0, 30, 45, 60, 90 and 120 min after consumption of protein supplements
Serum urea change from baseline | Blood collected at 0, 30, 45, 60, 90 and 120 min after consumption of protein supplements. For milk and native whey blood was collected at two additional time points: 22 and 30 hours after consumption of protein supplements
Muscle force generating capacity change from baseline | Measured before and at 0, 6, 22 and 30 hours after exercise. Only measured after milk and native whey
  Measured as unilateral isometric knee extension force (Nm) with 90° in the hip and knee joints.
Jump height change from baseline | Measured before and at 0, 6, 22 and 30 hours after exercise. Only measured after milk and native whey
  Measured as counter movement jump on a force plate
Serum creatine kinase change from baseline | Blood collected at 0, 30, 45, 60, 90 and 120 min after consumption of protein supplements. For milk and native whey blood was collected at two additional time points: 22 and 30 hours after consumption of protein supplements
Muscle soreness change from baseline | Measured before and at 0, 6, 22 and 30 hours after exercise. Only measured after milk and native whey
  Measured for m. quadriceps and m. pectoralis major on a visual analog pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Truls Raastad, PhD, Principal Investigator — Norwegian School of Sport Sciences

IPD SHARING:
Plan to Share IPD: Undecided